CLINICAL TRIAL: NCT07227753
Title: The Association Between Gut Microbiota Diversity and Postpartum Depression： A Prospective Pilot Study
Brief Title: The Association Between Gut Microbiota Diversity and Postpartum Depression
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jingping Wang, MD, Ph.D., Associate Professor, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2025P002566; 5R21AG081763 (NIH)
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Depression During Pregnancy
Keywords: depression; postpartum
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood (~5 mL; processed to serum and plasma) and rectal swab specimens will be collected around the time of delivery (pre-delivery within 3 days and early postpartum within 2 days). Specimens will be coded, stored at -80 °C, and used for laboratory analyses approved by the Institutional Review Board. No direct identifiers accompany specimens. No human whole-genome sequencing is planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-Edinburgh Postnatal Depression Scale cohort: Pregnant participants with antepartum Edinburgh Postnatal Depression Scale (EPDS; range 0-30; higher scores indicate more depressive symptoms) ≥13. Peripheral venous blood (serum) and rectal swab collected ≤3 days pre-delivery and ≤2 days postpartum; optional 6-week follow-up. Observational only-no interventions assigned.
- Low-Edinburgh Postnatal Depression Scale cohort: Pregnant individuals with antepartum Edinburgh Postnatal Depression Scale (EPDS; range 0-30; higher scores indicate more depressive symptoms) <13; same specimen collection and follow-up schedule as the high-EPDS cohort; no interventions assigned.

SUMMARY:
This study aims to examine whether naturally occurring bacteria in the gastrointestinal tract are associated with mood changes following childbirth, including postpartum depression. Biological samples will be collected before and after delivery to determine whether specific patterns in gut bacterial composition are linked to emotional states. The purpose of the research is to improve understanding of whether such microbial changes can help identify individuals at higher risk for postpartum depression, enabling earlier recognition and intervention.

DETAILED DESCRIPTION:
This prospective observational pilot study is designed to explore the relationship between gut microbial diversity and depressive symptoms during the early postpartum period. Postpartum depression is one of the most frequent complications after childbirth and has a substantial impact on the physical and psychological well-being of mothers and infants. The study investigates whether differences in gut microbial composition are associated with the development of depressive symptoms following childbirth.

Pregnant individuals aged eighteen years or older planning cesarean delivery at Massachusetts General Hospital will be enrolled. Data and biological samples will be collected at two time points: within three days before delivery and within 2 days after delivery. Blood samples will be collected for measurement of inflammatory markers, and rectal swab samples will be obtained to evaluate the composition and diversity of gut microorganisms through metagenomic sequencing. A validated questionnaire assessing emotional state will be administered at the same time points, and a follow-up emotional assessment will be obtained six weeks after childbirth through the electronic medical record system.

The study examines microbial characteristics associated with the presence or absence of depressive symptoms and evaluates correlations between microbial community patterns and emotional status, aiming to identify potential microbiome-based biomarkers predictive of early onset depressive symptoms after childbirth. The research does not include drug administration, device testing, or experimental treatment. All procedures are non-invasive or minimally invasive and coincide with routine obstetric care, minimizing participant burden.

The results of this study are expected to provide preliminary evidence linking the gut microbial environment to maternal mental health. Findings may inform future strategies for early detection and prevention of postpartum depressive symptoms and support the development of personalized approaches to maternal mental wellness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Gestational age at least 36 weeks, planned cesarean delivery
* Ability to understand study procedures and provide informed consent
* Voluntary agreement to participate in the study

Exclusion Criteria:

* Gastrointestinal disorders or recent antibiotic use that significantly alters gut microbiome
* Diagnosis of severe mental illness such as schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder with psychotic features
* Medication use during pregnancy known to influence gut microbiota, including antidepressants, antibiotics, or fish oil
* Refusal to provide rectal swab samples or inability to complete follow-up assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants are cisgender women who are pregnant or postpartum. Participants must have been assigned female at birth and currently self-identify as women.
Study Population: Women aged 18 years or older, with gestational age of at least 36 weeks, planning either vaginal or cesarean delivery. Individuals with serious digestive disorders, severe mental health conditions, or recent use of medications such as antibiotics or antidepressants that may affect gut bacteria are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
gut microbiota composition | within 3 days before delivery； within 2 days after delivery
  Compare gut microbiota composition between participants with postpartum depression (defined as Edinburgh Postnatal Depression Scale (EPDS; range 0-30; higher scores indicate more depressive symptoms) ≥13) and without postpartum depression (EPDS <13).

SECONDARY OUTCOMES:
Association between inflammatory cytokines and postpartum depressive symptom severity | Within 3 days before delivery; within 2 days after delivery
  Association between serum inflammatory cytokines (e.g., Interleukin-6, Tumor Necrosis Factor-alpha) and depressive symptom severity measured by the Edinburgh Postnatal Depression Scale (EPDS; range 0-30; higher scores indicate more depressive symptoms).
Edinburgh Postnatal Depression Scale (EPDS; range 0-30; higher scores indicate more depressive symptoms) | within 3days before delivery ; within 2 days after delivery; 6 weeks postpartum;
  Edinburgh Postnatal Depression Scale (EPDS; range 0-30; higher scores indicate more depressive symptoms) will be administered within 3 days before delivery ; within 2 days after delivery; 6 weeks postpartum;
Changes in gut microbiota diversity (alpha and beta) | within 3days before delivery ; within 2 days after delivery
  Alpha diversity (e.g., Shannon, Simpson, observed ASVs) and beta diversity (e.g., Bray-Curtis, UniFrac) will be calculated from rectal swab profiles. Change over time will be compared within participants.
Correlation between relative abundance of selected microbial taxa and maternal depressive symptom severity measured by the Edinburgh Postnatal Depression Scale (EPDS) | within 3days before delivery ; within 2 days after delivery
  Association between the relative abundance of prespecified taxa (e.g., Lactobacillus, Clostridium) from rectal swabs and Edinburgh Postnatal Depression Scale (EPDS; 0-30, higher scores indicate more depressive symptoms) at each timepoint and longitudinally within participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Meikun Wang, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. The dataset contains sensitive clinical information from pregnant and postpartum patients at a single institution.

REFERENCES:
- [Background] Sun Y, Fan C, Lei D. Association between gut microbiota and postpartum depression: A bidirectional Mendelian randomization study. J Affect Disord. 2024 Oct 1;362:615-622. doi: 10.1016/j.jad.2024.07.057. Epub 2024 Jul 17. PMID 39029663
- [Background] Bevilacqua G. [Prevention of perinatal infection caused by group B beta-hemolytic streptococcus]. Acta Biomed Ateneo Parmense. 1999;70(5-6):87-94. Italian. PMID 11402819
- [Background] Binka FN, Mensah OA, Mills A. The cost-effectiveness of permethrin impregnated bednets in preventing child mortality in Kassena-Nankana district of Northern Ghana. Health Policy. 1997 Sep;41(3):229-39. doi: 10.1016/s0168-8510(97)00035-3. PMID 10170091